CLINICAL TRIAL: NCT06613984
Title: Korean Post Marketing Surveillance for Comirnaty Injection
Brief Title: Korean Post Marketing Surveillance for Comirnaty Injection (Bretovameran)
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591072
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Vaccination
Keywords: COVID-19; Bretovameran; Adverse Events; SARS-Cov-2; Safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bretovameran: Korean subjects who are eligible for administration of Comirnaty Injection (Bretovameran) according to the locally authorized label
  Interventions: Biological: Bretovameran

INTERVENTIONS:
Biological: Bretovameran — Comirnaty Injection (Bretovameran) is administered intramuscularly as a single dose of 0.3 mL for individuals 12 years of age and older regardless of prior COVID-19 vaccination status.

SUMMARY:
This study is to identify any problems and questions with respect to the safety of Comirnaty Injection (Bretovameran) during the post-marketing period.

DETAILED DESCRIPTION:
All assessments are performed as part of normal clinical practice or standard practice guidelines for the subject population and healthcare provider specialty in the countries where this non-interventional study is being conducted.

This study is conducted under normal clinical practice in accordance with regulatory requirements. Therefore, the inclusion and exclusion criteria for study subjects are related to indications and contraindications outlined in the local product document. This study will not provide or make recommendations on any vaccine use. The vaccines are all given as part of the standard of care. All enrolled subjects have to meet the general prescription criteria for Comirnaty Injection (Bretovameran) according to the local product document and have to be enrolled at the doctor's discretion.

This is an open-label, non-comparative, non-interventional, prospective, and multi-center study conducted in Korean health care centers by accredited physicians (investigator). The study population is Korean subjects who are scheduled for COVID-19 vaccination. Comirnaty Injection (Bretovameran) will be administered according to the "Dosage and Administration" of the authorized label. There is no visit or activity mandated by this study. The investigator will collect data from the subject's medical records and diary and record data on each subject's case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Korean subjects who are eligible for administration of Comirnaty Injection according to the locally authorized label
* Subjects with evidence of a personally signed and dated informed consent/assent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Subjects who involved in the contraindications of use indicated in the locally authorized label
* Subjects with a history of hypersensitivity to any ingredients of this product or this product
* Any subjects (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is Korean subjects who are eligible for "indications" specified in the approved label.
  [INDICATIONS] Active immunisation to prevent COVID-19 caused by SARS-CoV-2, in individuals 12 years of age and older.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Solicited adverse events | 1 week after administration of Comirnaty Injection (Bretovameran)
  Solicited adverse events within 1 week after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Unsolicited adverse events | 28 days after administration of Comirnaty Injection (Bretovameran)
  Unsolicited adverse events within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.

SECONDARY OUTCOMES:
Number of subjects with Adverse events (AEs) | 28 days after administration of Comirnaty Injection (Bretovameran)
  All adverse events within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Serious Adverse Events (SAEs) | 28 days after administration of Comirnaty Injection (Bretovameran)
  All Serious adverse events within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Expected Adverse Events | 28 days after administration of Comirnaty Injection (Bretovameran)
  All expected adverse events within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Unexpected Adverse Events | 28 days after administration of Comirnaty Injection (Bretovameran)
  All Unexpected Adverse Events within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Adverse Drug Reactions | 28 days after administration of Comirnaty Injection (Bretovameran)
  All Adverse Drug Reactions within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Serious Adverse Drug Reactions | 28 days after administration of Comirnaty Injection (Bretovameran)
  All Serious Adverse Drug Reactions within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Expected Adverse Drug Reactions | 28 days after administration of Comirnaty Injection (Bretovameran)
  All Expected Adverse Drug Reactions within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.
Number of subjects with Unexpected Adverse Drug Reactions | 28 days after administration of Comirnaty Injection (Bretovameran)
  All Unexpected Adverse Drug Reactions within 28 days after each dose of Comirnaty Injection (Bretovameran) and the number of subjects with such events will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591072